CLINICAL TRIAL: NCT02775097
Title: Evaluation of the Accuracy of Corneal Epithelial Thickness Mapping With SD-OCT
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-50996
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-05

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Not having any history of refractive surgery, contact lens, dry eye or pathology
  Interventions: Device: OCT
- Corneal condition: History of refractive surgery, contact lens, dry eye or keratoconus.
  Interventions: Device: OCT

INTERVENTIONS:
Device: OCT — OCT for all Arms

SUMMARY:
Evaluate the accuracy of the RTVue-XR and iVue for measuring the total corneal thickness, the epithelial thickness, and the stromal thickness in normal subjects and patients with various corneal conditions.

ELIGIBILITY:
Inclusion Criteria:

Normal

* Able and willing to provide consent.
* Able and willing to complete required exams.

Corneal conditions

* Able and willing to provide consent.
* Able and willing to complete required exams.
* History of refractive surgery, contact lens, dry eye or keratoconus.

Exclusion Criteria:

Normal

* History of refractive surgery, contact lens, dry eye or pathology.
* Blepharitis or meibomitis
* Unable to complete required exams.

Corneal conditions

• Unable to complete required exams.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Epithelial thickness | Day 1

SECONDARY OUTCOMES:
Corneal thickness | Day 1

OTHER OUTCOMES:
Stromal thickness | Day 1